CLINICAL TRIAL: NCT03844269
Title: A Study to Assess Midline Frontal Theta (MFT) Power as Measured by Stimulus-locked Electroencephalography (EEG) Before and After AKL-T01 Treatment for Improving Attention in Pediatric Participants Ages 8-12 Years Old With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Electroencephalogram (EEG) Study of Inattention Following Treatment With AKL-T01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akili Interactive Labs, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 001S-C
Record Dates: First submitted 2019-02-14; First posted 2019-02-18 (Actual); Results first posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-10

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Inattention
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Intervention group will be compared to historical controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- AKL-T01 (Experimental)
  Interventions: Device: AKL-T01

INTERVENTIONS:
Device: AKL-T01 — AKL-T01 digital treatment is a state-of-the-art mobile video game-like platform, which deploys modern videogame graphics, engaging reward loops, and real-time adaptive mechanics to dynamically personalize difficulty based on the user's ability. AKL-T01 multitasking treatment employs perceptual discrimination attention/memory task as well as a continuous motor "driving" task. Performance on these tasks are assessed in isolation and when performed together to calculate a performance index for each individual user. A personalized multitask treatment regimen is automatically configured and delivered to the user and is optimized adaptively to increase multitask performance. As players proceed through the treatment periodic recalibration occurs to maintain an optimal difficulty level.

SUMMARY:
This study is a single arm, open-label, pilot study to assess midline frontal theta (MFT) power as measured by stimulus-locked electroencephalogram (EEG) before and after treatment with AKL-T01 for improving attention in pediatric participants ages 8-12 years old with attention deficit hyperactivity disorder (ADHD).

DETAILED DESCRIPTION:
All participants enrolled in this study will not be taking medications for attention deficit hyperactivity disorder (ADHD), including stimulants, for the duration of the study. Participants who are taking ADHD medications prior to Day 0 must have been stable off of medications for at least 30 days per parent report, or washout of medications at a Screening visit 3 - 7 days prior to Day 0.

At Baseline / Day 0, all eligible participants will complete both resting-state electroencephalogram (EEG) and a perceptual discrimination task (PDT)-locked EEG.

All participants will then play AKL-T01 for approximately 25 minutes per day, 5 days per week, for 4 weeks at home.

At Follow-up / Day 28, participants will repeat both resting-state and PDT-locked EEG.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed Attention Deficit Hyperactivity Disorder (ADHD) diagnosis at screening/baseline visit based on Diagnostic Diagnostic and Statistical Manual of Mental Disorders 5th Edition (DSM-V) criteria and established via the Mini-International Neuropsychiatric Interview for Children and Adolescents (MINI-KID) administered by a trained clinician either in person or via teleconference
* Wechsler Intelligence Scale for Children 5th Edition (WISC-V), Full Scale Intelligence Quotient ≥ 70
* Vanderbilt ADHD Diagnostic Parent Rating Scale: Must score a 2 or 3 on at least 6 items 1-9 AND must score a 4 on at least 2, or 5 on at least 1, of items 48-54 (performance questions).
* Consistently off stimulant medication for ≥ 1 week. OR currently on stimulant medication and agree to stop taking the medication for a 1 week prior to the baseline visit and off through duration of training and post-training assessment (note: participants will only be allowed to washout of stimulant medication if in the opinion of the investigator they are currently inadequately managed on their medication and it is appropriate to stop taking their medication for the duration of the trial)
* Consistently off Psychotropic drug for ≥ 1 month
* Consistently off non-stimulant medication for ADHD (e.g. atomoxetine, clonidine, guanfacine) for ≥ 1 month
* Able to follow written and verbal instructions (English) as assessed by the PI and/or study coordinator
* Functioning at an age-appropriate level intellectually
* Able to comply with all testing and requirements

Exclusion Criteria:

* Current controlled (requiring a restricted medication) or uncontrolled, comorbid psychiatric diagnosis, based on the Neurodevelopment Intake Form, Behavior Assessment System for Children (BASC), and subsequent clinical interviewing, with significant symptoms including but not limited to post-traumatic stress disorder, psychosis, bipolar illness, severe obsessive compulsive disorder, severe depressive or anxiety disorder, conduct disorder, or other symptomatic manifestations that in the opinion of the Investigator may confound study data/assessments. (Participants with clinical history of learning disorders will be allowed to participate as long as the disorder does not impact their ability to participate based on PI judgement).
* Autism Spectrum Disorder concern as indicated from the Social Communication Questionnaire ≥ 15.
* Current treatment with stimulant treatment for ADHD and unwilling or inappropriate (per investigator opinion) to washout.
* Initiation or completion of behavioral therapy within the last 4 weeks. The participant should inform the Investigator if they intend to change their behavioral therapy during the 4 weeks of the study. Participants who have been in behavior therapy consistently for more than 4 weeks may participate if their routine is unchanged throughout the study.
* Participant is currently considered at risk for attempting suicide by the Investigator, has previously made a suicide attempt, or has a prior history of, or is currently demonstrating active suicidal ideation or self-injurious behavior, as measured by MINI-KID Suicidality Module C.
* Motor condition (e.g. physical deformity of the hands/arms) that prevents game playing as reported by the parent or observed by the Investigator.
* Recent history or suspicion (within the past 6 months) of substance abuse or dependence.
* History of seizures (excluding febrile seizures).
* Participation in a clinical trial within 90 days prior to screening.
* Color blindness as detected by Ishihara Color Blindness Test.
* Regular use of psychoactive drugs that in the opinion of the Investigator may confound study data/assessments.
* Any other medical condition that in the opinion of the Investigator may confound study data/assessments.
* Previously received AKL-T01 (Project-EVO™) treatment in a previous clinical trial.
* Concurrent brain training

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2019-05-10 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elysa J Marco, MD, Principal Investigator — Cortica Healthcare
Locations (1):
- Cortica Healthcare, San Rafael, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gallen CL, Anguera JA, Gerdes MR, Simon AJ, Canadas E, Marco EJ. Enhancing neural markers of attention in children with ADHD using a digital therapeutic. PLoS One. 2021 Dec 31;16(12):e0261981. doi: 10.1371/journal.pone.0261981. eCollection 2021. PMID 34972140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AKL-T01
Started | 28
Completed | 25
Not Completed | 3
Not completed — Withdrawal pre-intervention | 1
Not completed — Did not complete the intervention | 2

BASELINE CHARACTERISTICS:
Arm/Group | AKL-T01
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.44 (1.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Midline Frontal Theta Power (MFT)
Description: Change in midline frontal theta (MFT) power as measured by Perceptual Discrimination Task (PDT)-Locked Electroencephalogram (EEG).
Time Frame: Day 0 to Day 28
Population: Exclusions: data with excessive noise at the pre- or post-intervention assessment. Excessive noise was defined as rejection of more than 30% of target trials due to voltage fluctuations greater than ± 100 μV deflections within an epoch.
Measure: Mean (Standard Deviation); unit: Hertz
Arm/Group | AKL-T01
Number analyzed (Participants) | 22
Hertz
  Mean change in time window 0-120 ms | -0.31835 (0.54423)
  Mean change in time window 160-280 ms | -0.15256 (0.79222)
  Mean change in time window 760-875 ms | -0.29013 (0.64112)
Statistical Analysis 1: Comparison: AKL-T01; EEG data excluded if excessive noise (rejection of more than 30% of target trials due to voltage fluctuations greater than ± 100 μV deflections within an epoch) at the pre- or post-intervention assessment; Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Midline Frontal Theta Power (MFT)
Description: MFT power as measured by Perceptual Discrimination Task (PDT)-Locked Electroencephalogram (EEG) of ADHD cohort post-treatment with AKL-T01 compared to that of neurotypical cohort at Day 0 (historical controls).
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hertz
Groups:
- Cortica Cohort: Participants enrolled in the present study, "Electroencephalogram (EEG) Study of Inattention Following Treatment with AKL-T01," with diagnosis of ADHD. All participants underwent 4-weeks of treatment with AKL-T01.
  Same as the "AKL-T01" group under Primary Outcome.
- Neurotypical Historical Control: EEG data from neurotypical participants from a prior study, "A pilot study to determine the feasibility of enhancing cognitive abilities in children with sensory processing dysfunction" (Anguera, 2017) was used as historical controls. All participants underwent 4-weeks of treatment with AKL-T01.
Arm/Group | Cortica Cohort | Neurotypical Historical Control
Number analyzed (Participants) | 22 | 18
Hertz
  Pre-intervention Mean MFT power (0-120 ms): number analyzed (Participants) | 21 | 18
  Pre-intervention Mean MFT power (0-120 ms) | .09047 (.625799) | -.34779 (1.278674)
  Post-intervention Mean MFT power (0-120 ms): number analyzed (Participants) | 21 | 18
  Post-intervention Mean MFT power (0-120 ms) | .39812 (.411608) | -.11458 (1.1151529)
  Pre-intervention Mean MFT power (200-320 ms): number analyzed (Participants) | 21 | 18
  Pre-intervention Mean MFT power (200-320 ms) | .81225 (.931336) | .54878 (2.391647)
  Post-intervention Mean MFT power (200-320 ms): number analyzed (Participants) | 21 | 18
  Post-intervention Mean MFT power (200-320 ms) | 1.06766 (.729074) | 1.09948 (1.804712)
  Pre-intervention Mean MFT power (680-800 ms): number analyzed (Participants) | 21 | 18
  Pre-intervention Mean MFT power (680-800 ms) | -.02013 (.436377) | -.05245 (2.444086)
  Post-intervention Mean MFT power (680-800 ms): number analyzed (Participants) | 21 | 18
  Post-intervention Mean MFT power (680-800 ms) | .35505 (.607502) | -.58763 (1.678055)

ADVERSE EVENTS:
Time Frame: 28 (+3) days
Description: No serious adverse events or mortality occurred during this trial.
Arm/Group | AKL-T01
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 0/28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT03844269/Prot_SAP_000.pdf